CLINICAL TRIAL: NCT00113360
Title: Phase II Study of RAD001 Plus Octreotide Depot in Patients With Metastatic or Unresectable Low Grade Neuroendocrine Carcinoma (Carcinoid, Islet Cell)
Brief Title: RAD001 Plus Octreotide Depot in Metastatic or Unresectable Low Grade Neuroendocrine Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2004-0597
Record Dates: First submitted 2005-06-07; First posted 2005-06-08 (Estimated); Results first posted 2010-12-07 (Estimated); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Neuroendocrine Carcinoma; Islet Cell Carcinoma
Keywords: Neuroendocrine Carcinoma; Low Grade Neuroendocrine Carcinoma; Neuroendocrine Carcinoid; Islet Cell Carcinoma; RAD001; Everolimus; Octreotide Depot; Sandostatin LAR; Octreotide long-acting release (LAR); Octreotide LAR
MeSH Terms: conditions — Carcinoma, Neuroendocrine; Carcinoma, Islet Cell | interventions — Everolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- RAD001 plus Depot Octreotide (Experimental): RAD001 at 5 or 10 milligrams orally once a day plus Octreotide Depot 30 milligrams intramuscularly once every 28 days.
  Interventions: Drug: RAD001; Drug: Octreotide Depot

INTERVENTIONS:
Drug: RAD001 — Starting dose of 5 or 10 mg by mouth daily.
  Other Names: Everolimus
Drug: Octreotide Depot — 30 mg injection into the muscle of either buttock once every 28 (±7) days.
  Other Names: Sandostatin LAR; Octreotide long-acting release (LAR); Octreotide LAR

SUMMARY:
Objectives:

Primary endpoint:

-Assess the clinical activity of RAD 001 plus depot octreotide as defined by progression free survival (PFS) duration defined by RECIST criteria in treated and untreated patients with metastatic, unresectable low grade neuroendocrine carcinoma.

Secondary endpoints:

* Assess the progression free survival duration of patients with metastatic, unresectable low grade neuroendocrine carcinoma treated with RAD 001 plus depot octreotide.
* Assess the safety of RAD 001 plus depot octreotide in patients with metastatic, unresectable low grade neuroendocrine carcinoma.
* To determine the expression/phosphorylation status of the components of the mTOR signaling pathway in the primary tumors, in order to determine whether these markers can be used as predictors of sensitivity to the combination of RAD001 and octreotide.
* To determine the effect of the combination of RAD001 and octreotide on the expression and phosphorylation of mTOR's targets in the accessible tumor tissue, in order to identify potential pharmacodynamics markers of response to this drug combination.
* To observe the effects of treatment with RAD001 on plasma angiogenic biomarkers.

DETAILED DESCRIPTION:
RAD001 is a new drug that is designed to block a protein that is important in the growth of cancer cells. Octreotide Depot is FDA approved for the treatment of carcinoid syndrome and hormonal symptoms from certain islet cell carcinomas. Octreotide Depot may also help to block certain proteins that are important in tumor growth.

Before you can start treatment on the study, you will have what are called "screening tests". These tests will help the doctor decide if you are eligible to take part in the study. You will be asked questions about your medical history and about any medications you are currently taking or have taken in the past. You will have a complete physical exam and your heart rate, temperature, breathing rate, blood pressure, height, and weight will be measured. You will be asked about your ability to perform every day activities. Blood (about 2 teaspoons) will be collected for routine tests. You will have an electrocardiogram (ECG - a test that measures the electrical activity of the heart) and scans (either Computed Tomography/CT or Magnetic Resonance Imaging/MRI) to evaluate the cancer. Women who are able to have children must have a negative blood pregnancy test.

If the screening evaluations show you are eligible to take part in the study, you may begin treatment. You will take RAD001 by mouth once a day, every day while on study. You should take it in a fasting state or after no more than a light, fat-free meal. You should take RAD001 about the same time each day. Octreotide Depot will be given as an injection into the muscle of either buttock once every 4 weeks while on study. This will be done at M. D. Anderson. Four weeks (28 days) is called one course of treatment.

Clinic visits will occur every 2 weeks during the first 4 weeks and every 4 weeks from then on. At each clinic visit, you will be asked questions about your medical history and about any medications you are currently taking or have taken in the past. You will have a complete physical exam and your heart rate, temperature, breathing rate, blood pressure, height, and weight will be measured. You will be asked about your ability to perform every day activities. Blood samples (about 1 teaspoons) for routine tests will be collected every 2 weeks for the first 8 weeks. After that, blood samples (about 2 teaspoons) will be collected every 4 weeks. CT or MRI scan(s) will be performed every 12 weeks.

If a sample of your tumor tissue that was removed previously is available, it will be analyzed for expression of proteins that may effect tumor growth. However, if a sample is not available, you will not be asked to undergo a biopsy to collect this tissue. This sample may analyzed at any time during the study.

If you experience severe side effects, treatment may be delayed, stopped, or you may receive smaller doses of RAD001 and/or Octreotide Depot. You may continue to receive up to at least 12 courses of study treatment unless the disease gets worse, you decide not to take part any longer, or your doctor decides it is in your best interest to stop treatment. It may be possible to continue treatment beyond 12 courses if you are benefitting from this treatment.

When you stop study treatment, you will be asked to have some tests and evaluations done. About 4 teaspoons of blood will be taken for routine lab tests, You will also have a physical exam and CT scan or MRI scan will be done to check the size and location of your disease.

This is an investigational study. RAD001 is investigational and is not commercially available. The drug combination in this study is also investigational. RAD001 is manufactured by Novartis Pharmaceuticals Corporation. About 60 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologic proof of low grade neuroendocrine carcinoma will be eligible. Both carcinoid (any site[atypical/intermediate grade carcinoid is allowed]) and islet cell (pancreatic endocrine tumor) will be eligible.
* Patients with neuroendocrine tumors associated with MEN1 syndrome will be eligible.
* Patients must have either metastatic or unresectable local-regional cancer.
* Patients must have measurable disease, as defined by RECIST (Response Evaluation Criteria In Solid Tumors).
* Prior and concurrent octreotide (Sandostatin and Sandostatin LAR) is allowed.
* Prior radiation therapy is permitted. A recovery period of at least 4 weeks after completion of radiotherapy is required prior to enrollment.
* Patients may have received 0, 1, or 2 prior cytotoxic chemotherapy.
* Chemotherapy used as a radiosensitizer will be considered one prior chemotherapy regimen.
* Patients may have received prior interferon (not counted toward prior cytotoxic chemotherapy).
* Patients may have received prior therapy targeting c-kit, abl, PDGFR (Platelet Derived Growth Factor Receptor), VEGF (Vascular endothelial growth factor), or EGFR [epidermal growth factor receptor] (not counted toward prior cytotoxic chemotherapy).
* Patients may have had prior hepatic artery embolization. There must be residual measurable disease. Chemoembolization will be considered as one prior chemotherapy regimen.
* Patients must have a performance status of 0, 1, or 2 (Zubrod scale).
* Patients must be >/= 18 years old (age limit due to lack of adequate safety data in younger patients).
* Patients must give written informed consent.
* Patients should have adequate organ function defined as follows: Absolute granulocytes > 1,500/mm3, hemoglobin > 8 g/dl, and platelets > 100,000/mm3. Serum bilirubin < 1.5 x Upper Limit of Normal (ULN), serum creatinine < 1.5 mg/dL, AST (SGOT) less/equal 2.5 x ULN, ALT (SGPT) less/equal 2.5 x ULN.
* Patients must have recovered from recent surgery. One week must have elapsed from the time of a minor surgery and 4 weeks from major surgery.
* Fertile patients, both male and female, must practice contraception during treatment.

Exclusion Criteria:

* Patients may receive no other concurrent chemotherapy, immunotherapy, or radiotherapy.
* Patients with intolerance to octreotide.
* Patients who have received chemotherapy, immunotherapy, or investigational therapy in the 30 days prior to registration.
* Patients with uncontrolled diabetes mellitus as defined by fasting blood sugar > 1.5 x ULN.
* Pregnant or lactating women. All women of child-bearing potential must have a negative pregnancy test prior to entry into the study. All patients of child-bearing potential must be advised of the importance of avoiding pregnancy and using appropriate methods of contraception while participating in this investigational trial. Women who have had menses within the past 2 years, who have not had a tubal ligation, or bilateral oophorectomy are considered to be of child-bearing potential. Appropriate methods of contraception include hormonal or barrier method of birth control; abstinence.
* Serious intercurrent infections, or nonmalignant medical illnesses that are uncontrolled or whose control may be jeopardized by the complications of this therapy.
* Psychiatric disorders rendering them incapable of complying with the requirements of the protocol.
* Osseous metastasis as only site of disease.
* Any concurrent active malignancy other than non-melanoma skin cancers or carcinoma-in-situ of the cervix. Patients with previous malignancies but without evidence of disease for > 5 years will be allowed to enter the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2005-01; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James Yao, M.D., Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center website — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment Period: 02/2005 to 07/2006. All participants were enrolled at UT M. D. Anderson Cancer Center.
Pre-assignment Details: Three subjects enrolled in the screening portion of the trial did not meet eligibility requirements based on laboratory measurements.
Groups:
- RAD001 Plus Octreotide Depot: RAD001 at 5 or 10 milligrams orally once a day plus Octreotide Depot 30 milligrams intramuscularly once every 28 days
Period: Overall Study
Arm/Group | RAD001 Plus Octreotide Depot
Started | 67 (67 participants were enrolled for screening.)
Completed | 60
Not Completed | 7
Not completed — Adverse Event | 3
Not completed — Subject required surgery | 1
Not completed — Did not meet eligibility criteria | 3

BASELINE CHARACTERISTICS:
Arm/Group | RAD001 Plus Octreotide Depot
Number analyzed (Participants) | 67
Age, Continuous [Mean (Full Range); unit: Years] | 55 [44 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36
  Male | 31
Region of Enrollment [Number; unit: participants]
  United States | 67

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS is measured from date of trial entry until documented progression of disease or death from any cause. PFS is measured by computed tomography (CT) scans or magnetic resonance imaging (MRI) performed at baseline and after every three cycles.
Time Frame: PFS assessed every 12 weeks (at the end of every 3 cycles) or more frequently if clinically indicated
Population: Per protocol
Measure: Median (95% Confidence Interval); unit: Weeks
Arm/Group | RAD001 Plus Octreotide Depot
Number analyzed (Participants) | 60
Weeks | 60 [54 to 66]

ADVERSE EVENTS:
Time Frame: 3 years, 6 months
Arm/Group | RAD001 Plus Octreotide Depot
Serious Adverse Events (participants affected / at risk) | 3/64
Other Adverse Events (participants affected / at risk) | 64/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RAD001 Plus Octreotide Depot (N=64)
Glucose, serum-high (hyperglycemia) (Investigations) | 1 (1)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hemoglobin (Blood and lymphatic system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | RAD001 Plus Octreotide Depot (N=64)
ALT, SGPT (Investigations) | 24 (37) — Alanine aminotransferase (ALT or SGPT)
AST,SGOT (Investigations) | 40 (51) — Aspartate aminotransferase (AST or SGOT)
Alkaline phosphatase (Investigations) | 6 (6)
Anorexia (Gastrointestinal disorders) | 4 (4)
Bilirubin (Investigations) | 4 (7)
Calcium, serum-low (hypocalcemia) (Investigations) | 4 (4)
Diarrhea (Gastrointestinal disorders) | 32 (73)
Dry skin (Skin and subcutaneous tissue disorders) | 6 (6)
Edema, limb (Blood and lymphatic system disorders) | 8 (11)
Fatigue (General disorders) | 40 (96)
Fever (in the absence of neutropenia) (General disorders) | 3 (3)
Flatulence (Gastrointestinal disorders) | 4 (4)
Glucose, serum-high (hyperglycemia) (Investigations) | 45 (76)
Glucose, serum-low (Hypoglycemia) (Metabolism and nutrition disorders) | 4 (5)
Hemoglobin (Blood and lymphatic system disorders) | 37 (43)
Injection site reaction (Skin and subcutaneous tissue disorders) | 30 (72)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 21 (42) — White Blood Count (WBC)
Magnesium, serum-low (Hypomagnesemia) (Metabolism and nutrition disorders) | 18 (21)
Mucositis/stomatitis (functional/symptomatic) (Gastrointestinal disorders) | 38 (149)
Nail changes (Skin and subcutaneous tissue disorders) | 6 (6)
Nausea (Gastrointestinal disorders) | 28 (63)
Neutrophils/granulocytes (ANC/AGC) (Blood and lymphatic system disorders) | 25 (40) — Absolute neutrophil count (ANC)/Absolute granulocytes count (AGC)
Pain (Abdomen NOS) (General disorders) | 4 (4) — Not otherwise specified (NOS)
Pain (Head/Headache (General disorders) | 17 (28)
Pain (other) (General disorders) | 4 (8)
Pain - Other (injection site) (General disorders) | 3 (3)
Pain-Other (Buttock) (General disorders) | 4 (5)
Phosphate, serum-low (Hypophosphatemia) (Investigations) | 20 (28)
Platelets (Blood and lymphatic system disorders) | 24 (41)
Pneumonitis/pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Potassium, serum-high (hyperkalemia) (Investigations) | 5 (5)
Potassium, serum-low (Hypokalemia) (Metabolism and nutrition disorders) | 10 (18)
Pruritus/itching (Skin and subcutaneous tissue disorders) | 4 (4)
Rash/desquamation (Skin and subcutaneous tissue disorders) | 22 (48)
Rash: Erythema multiforme (Skin and subcutaneous tissue disorders) | 8 (12)
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 12 (16)
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 16 (17)
Thyroid function, low (hypothyroidism) (Endocrine disorders) | 3 (3)
Triglyceride, serum-high (hypertriglyceridemia) (Investigations) | 29 (43)
Vomiting (Gastrointestinal disorders) | 8 (16)
Weight loss (General disorders) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No